CLINICAL TRIAL: NCT03656003
Title: A Study Evaluating the Diagnostic Yield and Safety of the ProCore vs Conventional EBUS-TBNA Needle in Subjects With Suspected Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Int/IEC/2018/00169
Record Dates: First submitted 2018-08-22; First posted 2018-09-04 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procore needle (Experimental): EchoTip ProCore needle (Cook Medical Inc., Bloomington, Ind., USA)
  Interventions: Device: Procore biopsy needle
- Conventional needle (Active Comparator): Conventional 22-gauge EBUS-TBNA needle (Vizishot, Olympus, Japan)
  Interventions: Device: Conventional biopsy needle

INTERVENTIONS:
Device: Procore biopsy needle — EBUS-TBNA with the EchoTip ProCore needle (Cook Medical Inc., Bloomington, Ind., USA)
  Arms: Procore needle
Device: Conventional biopsy needle — EBUS-TBNA with the conventional 22-gauge EBUS-TBNA needle (Vizishot, Olympus, Japan)
  Arms: Conventional needle

SUMMARY:
This study evaluates the yield and safety of two different needles for performing endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA) in patients with sarcoidosis. The two needles that will be compared will be the 22-gauge ProCore needle and the conventional 22-gauge EBUS-TBNA needle.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem disorder of unknown cause characterized by granulomatous inflammation involving various organ systems. The diagnosis is made on the basis of a suggestive clinicoradiological picture, histopathologic evidence of non-caseating granuloma, and exclusion of other known causes for granulomatous inflammation. As the lung and mediastinal lymph nodes are the most commonly involved structures in sarcoidosis, various bronchoscopic techniques like endobronchial biopsy (EBB), transbronchial biopsy (TBLB) and transbronchial needle aspiration (TBNA) are needed for tissue sampling.

Among the bronchoscopic techniques, TBNA of lymph nodes is a useful modality especially when combined with endobronchial and transbronchial biopsies. The efficacy and safety of conventional TBNA are well established. With the advent of endobronchial ultrasound (EBUS) in the last decade, this new technology has been widely used to guide transbronchial needle aspiration. The technique is minimally invasive and offers the additional advantage of choosing the appropriate node for sampling based on the vascularity, echogenicity and size. Studies subsequently have demonstrated the superiority of EBUS-TBNA over conventional TBNA.

As EBUS-TBNA is the standard procedure now for accessing intrathoracic lymph nodes, the technical aspects of the procedure need further investigation. Several aspects have been studied to optimize the yield including the number of aspirations or passes required per lymph node station, needle gauge (21 vs. 22 gauge), suction pressure, and the distance travelled by the needle within the lymph node.

The EchoTip ProCore High Definition ultrasound biopsy needle (Cook Medical Inc., Bloomington, Ind., USA) is a novel needle that has been used mainly in sampling intra-abdominal lesions. It has a special bevel which allows a core biopsy along with aspiration of the lymph node material. In case of mediastinal lymph node enlargement due to malignancy, needle aspiration alone may yield sufficient material to identify malignant cells. However, in sarcoidosis, the core biopsy specimen obtained with the ProCore needle may potentially increase the identification of granulomas. The investigators hypothesize that the 22-gauge ProCore needle will have a higher yield in diagnosing intrathoracic lymphadenopathy due to sarcoidosis as compared to the conventional 22-gauge EBUS-TBNA needle. In this study, the investigators plan to evaluate the yield and safety of the 22-gauge ProCore needle as compared to the conventional 22-gauge EBUS-TBNA needle in patients with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria: Patients meeting all the following criteria will be eligible for inclusion in the study:

* Age group of 18 to 75 years
* Clinicoradiological suspicion of sarcoidosis where EBUS-TBNA is being planned
* Enlarged hilar and mediastinal lymph nodes >10 mm (any axis) on computed tomography of the chest
* Ability to provide informed consent to participate in the study

Exclusion Criteria: Patients with any of the following will be excluded:

* Hypoxemia (SpO2 <92% on FiO2 of 0.3)
* Treatment with systemic glucocorticoids for >2 weeks in the preceding three months
* Diagnosis of sarcoidosis possible with another minimally invasive technique such as skin biopsy or peripheral lymph node biopsy
* Failure to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sarcoidosis diagnosed by EBUS-TBNA (Diagnostic yield) | 6 months
  The diagnostic yield is defined as the proportion of patients with a final diagnosis of sarcoidosis diagnosed by EBUS-TBNA

SECONDARY OUTCOMES:
Number of patients with adequate EBUS-TBNA aspirate on cytology | 2 weeks
  Defined as preponderance of lymphocytes or a definite diagnosis (sarcoidosis, tuberculosis or others) on EBUS-TBNA aspirate
Incidence of adverse events related to EBUS-TBNA procedure in the two groups | 1 week
  Endobronchial bleeding, pneumothorax, hypoxemia, mediastinitis

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh N Aggarwal, Study Chair — Professor & Head
Locations (1):
- Bronchoscopy suite, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhooria S, Sehgal IS, Prasad KT, Muthu V, Gupta N, Bal A, Ram B, Aggarwal AN, Agarwal R. Diagnostic yield and safety of the ProCore versus the standard EBUS-TBNA needle in subjects with suspected sarcoidosis. Expert Rev Med Devices. 2021 Feb;18(2):211-216. doi: 10.1080/17434440.2021.1876560. Epub 2021 Jan 22. PMID 33435733